CLINICAL TRIAL: NCT07258173
Title: Efficacy and Safety of a Single Dose of Emodepside Compared to a Single Dose of Albendazole in Adolescents and Adults Infected With Trichuris Incognita: a Phase II, Randomized, Double Blind, Controlled Trial
Brief Title: Efficacy and Safety of a Single Dose of Emodepside Compared to a Single Dose of Albendazole in Adolescents and Adults Infected With Trichuris Incognita
Acronym: EMOTI
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jennifer Keiser (Other)
Collaborators: Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other); Université Félix Houphouët-Boigny (Unknown); Bayer (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Keiser, Professor, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EMODEPSIDE_CÔTE_D'IVOIRE
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Trichuris Infection; Trichuris
Keywords: Trichuris incognita; emodepside; efficacy; safety; soil transmitted helminths; Trichuris; Côte d'Ivoire
MeSH Terms: conditions — Trichuriasis | interventions — emodepside; Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Emodepside 15mg (Experimental)
  Interventions: Drug: Emodepside
- Albendazole 400 mg (Active Comparator)
  Interventions: Drug: Albendazole 400 mg

INTERVENTIONS:
Drug: Emodepside — Treatment with 15 mg of emodepside
  Arms: Emodepside 15mg
Drug: Albendazole 400 mg — Treatment with 400mg of albendazole
  Arms: Albendazole 400 mg

SUMMARY:
The purpose of this clinical trial is to compare the efficacy and safety of emodepside, with the standard treatment, albendazole, in adolescents (12 years and older) and adults infected with Trichuris incognita.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12 years and above.
* Written informed consent signed by participant and, in the case of minors, parents/caregivers.
* Agree to comply with study procedures, including provision of two stool samples at the beginning (screening) and at follow-up assessment 14-21 days after treatment.
* Having at least two slides of the quadruple Kato-Katz thick smears positive for Trichuris incognita and infection intensities of at least 48 eggs per gram (EPG).
* Willing to be examined by a study physician prior to treatment.

Exclusion Criteria:

* Presence or signs of major systemic illnesses, e.g. body temperature ≥ 38 °C, severe anemia (Hb below 80g/l) upon initial clinical assessment etc.
* History of severe acute or unmanaged severe chronic disease (i.e., condition is not as therapeutically controlled as necessary).
* Positive malaria rapid diagnostic test (RDT) and temperature ≥ 38 °C.
* Abnormal liver and renal function assessed by biochemical blood-based analyses
* Recent use of anthelmintic drugs (in the 4 weeks before treatment).
* Known allergy to study medications and formulations (i.e., albendazole and emodepside).
* Prescribed or taking medication with known contraindication to or interaction with study drugs.
* Participating in other clinical trials during the study period.
* Pregnancy or breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Cure rate (CR) of emodepside compared to albendazole against Trichuris incognita | Between 14-21 days post-treatment
  Trichuris incognita infection status of participants 14-21 days post-treatment assessed by Kato-Katz. CRs will be calculated as the percentage of egg-positive participants at screening who become egg-negative after treatment, for each treatment arm. Differences in CRs between the two treatments will be assessed.

SECONDARY OUTCOMES:
Egg-reduction rate (ERR) of emodepside compared to albendazole against Trichuris incognita | Between 14-21 days post-treatment
  Eggs per gram of stool (EPG) will be assessed by adding up the egg counts from the quadruplicate Kato-Katz thick smears and multiplying this number by a factor of six. Geometric mean egg counts will be calculated for the different treatment arms before and after treatment to assess the corresponding ERRs. ERR is caluclated as follows: ERR = (1- (geometric mean EPG at follow-up ÷ geometric mean EPG at baseline)) x 100
Safety and tolerability | 3- and 24- hours post-treatment and retrospectively 14-21 days post-treatment
  Tolerability of treatments (adverse events (AEs)) will be assessed at 3- and 24- hours post-treatment and at 14 - 21 days follow up. The safety analysis will be conducted on all participants who were treated and include all available drug safety data. AEs will be evaluated descriptively as the difference between proportions of reported AEs before and after treatment.

OTHER OUTCOMES:
CR and ERR of emodepside and albendazole against Ascaris lumbricoides and hookworm in co-infected participants | Between 14-21 days post-treatment
  If there are enough co-infections in the sample, exploratory analyses will be performed to assess the difference in cure rates and ERR for hookworm and A. lumbricoides. If there are fewer than 30 participants with co-infections of a certain species in total, the results will only be provided descriptively.

IPD SHARING:
Plan to Share IPD: Undecided